CLINICAL TRIAL: NCT01516450
Title: An Open Label, Randomized, Parallel, Single Dose Study to Investigate Safety and Pharmacokinetics Following Intravenous Administration and Subcutaneous Administration of GSK1550188 in Healthy Japanese Males
Brief Title: Japanese phase1 Study of Belimumab (IV vs SC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 116119
Record Dates: First submitted 2011-12-21; First posted 2012-01-24 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: GSK1550188, belimumab, SLE, healthy, Japanese, pharmacokinetics, safety
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1550188 200mg for SC (Active Comparator): Single SC dose of belimumab 200mg
  Interventions: Drug: GSK1550188 SC
- GSK1550188 200mg for IV (Active Comparator): Single IV dose of belimumab 200 mg
  Interventions: Drug: GSK1550188 IV

INTERVENTIONS:
Drug: GSK1550188 IV — Single IV dose of belimumab 200 mg
  Arms: GSK1550188 200mg for IV
Drug: GSK1550188 SC — Single SC dose of belimumab 200mg
  Arms: GSK1550188 200mg for SC

SUMMARY:
This study is an open-label, randomized, 2 parallel group, single dose study in healthy Japanese males to assess the pharmacokinetics and safety/tolerability of single intravenous administration and single subcutaneous administration of GSK1550188. Serial blood samples for the determination of GSK1550188 concentration will be collected and safety assessments will be performed for each treatment group

ELIGIBILITY:
Inclusion Criteria:

* Healthy as defined as being free from clinically significant illness or disease as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital sign, laboratory tests and ECG. Rationale: Set for the appropriate selection of healthy males
* Japanese healthy male between 20 and 55 years of age inclusive, at the time of signing the informed consent. Rationale: Set for the appropriate evaluation of safety and pharmacokinetics of GSK1550188 in healthy Japanese males
* Body weight greater than and equal to 50.0 kg and BMI within the range 18.5 more than and equal to - less than 25.0 kg/m2. Rationale: To include those who have a standard figure based on the obesity criteria of the Obesity Association in Japan, these ranges are established
* Non-smoker or ex-smoker having ceased smoking for at least 6 months. Rationale: Set for the appropriate evaluation of safety and pharmacokinetics of GSK1550188 in healthy Japanese males
* AST, ALT, alkaline phosphatase and total bilirubin less than and equal to ULN at screening. Rationale: Set for the appropriate evaluation of safety and pharmacokinetics of GSK1550188 in healthy Japanese males
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. Rationale: Set in consideration of ethics of the study in accordance with GCP.
* Single QTc [QTcF] less than 450 msec. Rationale: Set for the appropriate evaluation of safety and pharmacokinetics of GSK1550188 in healthy Japanese males

Exclusion Criteria:

* A positive test for syphilis, Hepatitis B surface antigen, Hepatitis B surface antibody, Hepatitis B core antibody, or positive Hepatitis C antibody, HIV antigen /antibody, HTLV-1 antibody at screening. Rationale: Set for the appropriate selection of healthy subjects and in consideration of safety of the staff that handle or measure the blood samples.
* A positive pre-study drug screen at screening. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of regular alcohol consumption exceeding, on average, 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* The subject had participated in a clinical study or post-marketing study with an investigational or a non-investigational product during the previous 4 months preceding the administration of study medication of this study. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* Exposure to more than four new chemical entities within 12 months prior to the dosing day. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* The subject planned to concurrently participate in another clinical study or post-marketing study. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the administration of study medication. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy excluding pollen allergy without current symptoms. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* Where participation in the study would result in donation of blood or blood products in excess of 400 mL within 4 month or 200 mL within 2 months.
* Unwillingness or inability to follow the procedures outlined in the protocol. Rationale: Set to secure study quality
* Subject is mentally or legally incapacitated. Rationale: Set to secure study quality
* Subjects with ECG results considered clinically significant by the investigator. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* Subjects with a supine systolic blood pressure less than 90 mmHg or greater than140 mmHg and/or a supine diastolic blood pressure less than 55 mmHg or greater than 90 mmHg and/or systolic blood pressure drop from supine to standing of greater than 30 mmHg. Rationale: Set in consideration of subjects' safety related to the IV route of administration.
* Immunoglobulin (M, A, G) level is less than LLN at screening. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of anaphylactic reaction to any food, drug, or insect bite/sting. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of allergic reaction to parenteral administration of contrast agents, foreign proteins, or monoclonal antibodies. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of B cell targeted therapy (rituximab, other anti-CD20agents, anti-CD22 [epratuzumab], anti-CD52 [alemtuzumab], BLyS-receptor fusion protein [BR3], TACI-Fc, LY2127399 [anti-BAFF] or GSK1550188) at any time. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.
* History of any infection requiring hospitalization or treatment with antivirals or antibiotics, or vaccination within 30 days prior to administration of study medication. Rationale: To exclude inappropriate subjects for the evaluation of the safety and pharmacokinetics of GSK1550188.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12-26 (Actual); Primary Completion 2012-04-11 (Actual); Study Completion 2012-04-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Vital signs | Day1-Day71
  Systolic and diastolic blood pressure, pulse rate, body temperature
Change from baseline of biomarkers | Day-1 - Day71
  CD20+, immunoglobulin
Immunogenicity | Day0 - Day71 (if necessary, 6-month)
  Presence of anti belimumab antibody
Change from baseline of other safety parameters after single intravenous and subcutaneous administration | Day-1 - Day71
  ECGs, clinical laboratory test, local tolerance evaluation (injection site), and adverse events

SECONDARY OUTCOMES:
Composite (or profile) of pharmacokinetics after single intravenous administration | Day1-Day71
  Percentage of AUC(0-inifinity) obtained by extrapolation (%AUCex), Time of last quantifiable concentration (tlast), Systemic clearance of parent drug (CL), Volume of distribution after IV/SC administration (Vz), Volume of distribution after IV administration at steady state (Vss), Terminal phase rate constant (λz), Mean residence time(MRT)
Composite (or profile) of pharmacokinetics after subcutaneous administration | Day-1 - Day71
  Area under concentration-time curve (AUC) 0-7days, AUC 0-28 days, Percentage of AUC(0-infinity) obtained by extrapolationAUC(0-infinity) (%AUCex), tlast, Apparent clearance following subcutaneous dosing (CL/F), Volume of distribution after IV/SC administration (Vz)/F, λz, MRT

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Gupta SV, Fanget MC, MacLauchlin C, Clausen VA, Li J, Cloutier D, Shen L, Robbie GJ, Mogalian E. Clinical and Preclinical Single-Dose Pharmacokinetics of VIR-2218, an RNAi Therapeutic Targeting HBV Infection. Drugs R D. 2021 Dec;21(4):455-465. doi: 10.1007/s40268-021-00369-w. Epub 2021 Nov 6. PMID 34741731
- [Derived] Zhou X, Lee TI, Zhu M, Ma P. Prediction of Belimumab Pharmacokinetics in Chinese Pediatric Patients with Systemic Lupus Erythematosus. Drugs R D. 2021 Dec;21(4):407-417. doi: 10.1007/s40268-021-00363-2. Epub 2021 Oct 9. PMID 34628605
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116119 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116119?search=study&study_ids=116119#rs
- Available data/document: Clinical Study Report: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116119 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register